CLINICAL TRIAL: NCT03863756
Title: Contribution of EOS in the Structural Evaluation of Spondyloarthritis
Brief Title: Performance of EOS Imaging System in the Assessment of Spondyloarthritis Structural Changes Compared With Standard Radiography
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Faculty of Medicine of Tunis (Other)
Collaborators: Institut Kassab d'Orthopédie (Other)
Responsible Party: Principal Investigator, Hamdi Ons, principal investigator, Faculty of Medicine of Tunis
Other Study IDs: Institut d'orthopédie Kassab
Record Dates: First submitted 2019-03-03; First posted 2019-03-05 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Spondyloarthritis
Keywords: spondyloarthritis; spine; syndesmophyte; radiography; EOS
MeSH Terms: conditions — Spondylarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: EOS — The new EOS-technology (EOS imaging, Paris, France) based on a low-dose X-ray system allows 3D modeling of the spine based on 2-dimensional
  Other Names: Standard radiography

SUMMARY:
Spondyloarthritis is a chronic rheumatic disease that requires prolonged radiographic follow-up. This repetitive exposure to ionizing radiation puts at risk the radiosensitive organs exposed in the field of irradiation. A new low-dose imaging system has emerged. This technique, called EOS, offers the advantage of lower irradiation associated with high images quality. Our goal through this work was to evaluate the reliability of the EOS imaging system compared to conventional radiography in the evaluation of the structural damage of SpA.

DETAILED DESCRIPTION:
Spondyloarthritis (SpA) is a chronic inflammatory disease that can affect the sacroiliac joints, the spine and / or the peripheral joints. It is characterized by a progressive and slow evolution over several years with a risk of ankylosis of the spine. It requires long-term follow-up of patients with repeated x-rays to assess structural damage. This repeated and cumulative exposure to radiation ionization puts at risk the radiosensitive organs that are in the field of irradiation.

EOS is a new low dose X-ray system that significantly reduces X-ray doses compared to conventional radiography. This system allows the global assessment of the entire skeleton from head to toe, static spine and lower limbs with the obtaining of two-dimensional images of high quality with the possibility of a three-dimensional reconstruction. Although the benefits of the EOS system are promising with regard to radiation dose reduction, few studies have investigated its use in SpA and little evidence has supported its reliability in assessing the structural damage caused by the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Spondyloarthritis (SpA) meeting the criteria of Amor and / or Assessement of spondyloarthritis International Society (ASAS)
* Indication of standard radiography for the follow-up of the patients.

Exclusion Criteria:

* the presence of a contraindication to the performance of conventional radiography (CR) or EOS imaging
* any disease affecting cognition
* Patients who have had surgery on the spine and / or hip.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General data demographics , disease characteristics [symptom duration, disease presentation (axial/peripheral), SpA features (psoriasis, uveitis, Human Leukocyte Antigen(HLA) B27 positivity)], disease activity: Bath ankylosing spondylitis disease activity index ( BASDAI) and C-reactive protein (CRP) and disease severity:Bath Ankylosing Spondylitis Functional Index (BASFI) data were collected.
  CR technique: All patients underwent a posteroanterior pelvic CR and a lateral and anteroposterior CR of the full spine.
  EOS technique: all patients undewent a full spine and pelvis 2D EOS imaging.
Sampling Method: Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Intermodality agreement | 6 months
  measuring the intermodality agreement between EOS and conventional radiography for the assessment of both the sacro-iliac joints and the spine by using 3 scores: the modified New York criteria, the modified Stoke Ankylosing Spondylitis Spinal Score (mSASSS) and the Bath Ankylosing Spondylitis Radiology Index (BASRI).

SECONDARY OUTCOMES:
interreader agreement | 3 months
  measuring the interreader agreement between the radiologist and the rheumatologist for the assessement of the sacro-iliac joints and the spine

CONTACTS AND LOCATIONS:
Overall Officials: Mataallah Kaouther, university hospital lecturer, Study Director — Institut d'orthopédie Kassab; Riahi Hend, university hospital lecturer, Study Director — Institut d'orthopédie Kassab; Hamdi Wafa, University Hospital Professor, Study Chair — Institut d'orthopédie Kassab; Chelli Mouna, University Hospital Professor, Study Chair — Institut d'orthopédie Kassab; Kaffel Dhia, Associate professor, Study Chair — Institut d'orthopédie Kassab; Ferjani Hanene, university hospital lecturer, Study Chair — Institut d'orthopédie Kassab
Locations (1):
- Institut d'orthopédie Kassab, Tunis, Mannouba, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maatallah K, Hamdi O, Bouaziz M, Lassoued H, Labbene E, Ladeb F, Kaffel D, Riahi H, Hamdi W. EOS: A new tool with weaknesses for assessing structural changes in spondyloarthritis. Joint Bone Spine. 2022 Jul;89(4):105328. doi: 10.1016/j.jbspin.2021.105328. Epub 2021 Dec 11. No abstract available. PMID 34906697